CLINICAL TRIAL: NCT01219582
Title: Open, Prospective, Multicentric, Single-arm, Non-interventional Study to Evaluate the Effectiveness & Safety of Oral Glucobay®-M Tablets in Type 2 Diabetes Patient
Brief Title: GLucobay M OBservation Study for Efficacy and Safety in Treatment of Type-2 Diabetes Patients
Acronym: GLOBE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14954; GB0910IN (Other: company internal)
Record Dates: First submitted 2010-10-07; First posted 2010-10-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus Type-2; Acarbose; Metformin; Drug Therapy, Combination
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Glucobay M (Acarbose/Metformin, BAY81-9783)

INTERVENTIONS:
Drug: Glucobay M (Acarbose/Metformin, BAY81-9783) — Oral Glucobay-M 25 every 8 hours (Q8H) titrated to Glucobay-M 50 Q8H or as per investigators discretion.

SUMMARY:
An observational and multicenter study to assess the effectiveness and safety of Glucobay®- M under daily life treatment of type-2 diabetes patients.The study objectives are to investigate the effectiveness and safety of Glucobay® -M on blood glucose and patients body - weight. Glucobay®- M is taken 1-3 times daily. All patients with type 2 diabetes mellitus, where investigator feels that addition of Glucobay®-M would be beneficial to patients will be included in non- interventional study. The routine investigation suggested by the attending physician will be done in diabetic patients. No additional investigation will be done for the study purpose. The uncontrolled diabetic patient on existing treatment and prescribed Glucobay®-M will be included in study after taking the informed consent. The patient will be asked to attend 2 follow up visit each after 6 weeks. All patients receiving at least one tablet will be included in the safety analysis.The study is planned to be carried out in 10000 patients from 320-350 trial sites in India.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 18 years of age with Type 2 Diabetes where investigator feels that addition of Glucobay®-M would be beneficial to patients.
* The diagnosis will be made based on the ADA criteria by the attending physician.
* Patients will be defined as included in the study if they have a documented prescription of Glucobay-M by the physician.
* Patients willing to provide signed & dated informed consent.
* Patients willing to comply with study requirements.

Exclusion Criteria:

* According to the local product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetes
Sampling Method: Probability Sample
Enrollment: 9364 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in fasting blood glucose levels | 12 weeks
Change in post-prandial glucose values | 12 weeks
Change in Hemoglobin A1c (HbA1c) levels | 12 weeks

SECONDARY OUTCOMES:
Number of patient with adverse events | 12 weeks
Percentage of patients with satisfaction of treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, India